CLINICAL TRIAL: NCT06654739
Title: Randomized, Sham Controlled, Single Blind Study on the Performance and Safety of Photo Biomodulation Therapy (PBMT) With LightForce® Therapy Lasers on Knee Osteoarthritis Pain Reduction
Brief Title: RCT on the Performance and Safety of LightForce® Therapy Lasers on Knee Osteoarthritis Pain Reduction (SPARK)
Acronym: SPARK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DJO UK Ltd (Industry)
Collaborators: Donawa Lifescience Consulting SRL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENOVIS-S-INP-0001
Record Dates: First submitted 2024-10-18; First posted 2024-10-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Laser Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized, sham controlled, single blind
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment arm 1 (Sham Comparator): Sham laser therapy + standard of care (SOC) represented by physiotherapy/exercise protocol
  Interventions: Device: Sham Laser therapy + physiotherapy/exercise protocol
- Treatment arm 2 (Active Comparator): Laser therapy + standard of care (SOC) represented by physiotherapy/exercise protocol
  Interventions: Device: Laser therapy + physiotherapy/exercise protocol

INTERVENTIONS:
Device: Laser therapy + physiotherapy/exercise protocol — laser therapy + standard of care (SOC) represented by physiotherapy/exercise protocol (program includes kinesitherapy, range of motion (ROM) exercises, stretching, strengthening, and flexibility exercises) for 6 consecutive weeks, for a minimum of 2 sessions per week
  Arms: Treatment arm 2
Device: Sham Laser therapy + physiotherapy/exercise protocol — sham laser therapy + standard of care (SOC) represented by physiotherapy/exercise protocol (program includes kinesitherapy, range of motion (ROM) exercises, stretching, strengthening, and flexibility exercises) for 6 consecutive weeks, for a minimum of 2 sessions per week
  Arms: Treatment arm 1

SUMMARY:
DJO UK Ltd (ENOVIS) is conducting this study to assess the effectiveness of LightForce® Therapy Lasers on pain reduction in subjects with unilateral or bilateral knee osteoarthritis. In detail this study will assess superiority of LightForce® Therapy Lasers combined with standard of care, represented by physiotherapy/exercise program compared to sham laser combined with standard of care (physiotherapy/exercise program) on pain reduction in subjects with knee osteoarthritis. In addition, this study allows to collect post market clinical data on the safety and performance of LightForce® Therapy Lasers, when used, following the normal clinical practice, in accordance with its approved and CE marked intended use.

DETAILED DESCRIPTION:
This clinical investigation is a post-market, International, multi center, prospective, randomized, sham controlled, single blind study to assess the effectiveness of LightForce® Therapy Lasers and to collect PMCF data on the safety and performance of LightForce® Therapy Lasers, when used in accordance with its approved labeling, to comply with Medical Device Regulation (EU) 2017/745 (MDR) Article 61 and Part B of Annex XI.

ELIGIBILITY:
Inclusion Criteria:

* Patient male or female with age ≥18 years old
* Patient with radiographic diagnosis of knee osteoarthritis (as confirmed by x- ray or CT scan) to be treated by LightForce® Therapy Lasers according its indications.
* Patient with Kellgren and Lawrence grade 2-3 unilateral or bilateral knee osteoarthritis
* Patient suffering from knee osteoarthritis pain for more than 6 months prior to enrollment
* Pain (either persistent or during activities) score reported by the subject at baseline ≥ 40 mm measured on VAS
* Patient able to provide written informed consent
* Patient with BMI ≤30 kg/m2
* For FRANCE ONLY: To be affiliated to the social security system or to be beneficiary of such system

Exclusion Criteria:

* Patient with musculoskeletal pathological conditions not to be treated with/contraindication to the use of LightForce® Therapy Lasers according to its intended use and indications
* Patients who are taking drugs that have heat or light sensitive contraindications, such as but not limited to certain types of steroids
* Patients who are administered with corticosteroids, should discontinue the treatment at least 2 weeks prior to study treatment start
* Pregnant females or females of childbearing potentially planning to become pregnant during the study participation
* Patients who had inflammatory arthritis (i.e. rheumatoid arthritis, psoriatic arthritis)
* Patients who underwent intra-articular injection (Ialuronic acid, platelet rich plasma or corticosteroids) in the knee in the last 6 months
* Patients who have a disease that would limit their participation in exercises (i.e. severe chronic obstructive pulmonary disease, severe heart failure, cerebrovascular event history)
* Patients who have hip or ankle/foot joint pathology that might interfere with participation in exercises/knee recovery
* Patients with a diagnosis of active cancer
* Patients with tattoos covering more than 30% of the area to be treated with LightForce® Therapy Lasers
* Patients who are mentally or physically incapacitated
* Patient participating in other clinical study or has completed a clinical study less than 30 days prior to enrollment
* Patients with other musculoskeletal problems of the knee joint such as tendon or ligament injury, recent surgery, recent fracture, or recent meniscus injury and/or undergoing to specific physiotherapy for these ("recent" is defined as within 30 days prior to enrollment)
* Patients with other clinically significant co-morbidities that make the patient unsuitable for study participation, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-11-23 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain change | 6 weeks after treatment start
  Pain reduction measured with Visual Analog Scale (VAS) (0-100 mm) after 6 weeks of treatment compared to pre-treatment (baseline) VAS

SECONDARY OUTCOMES:
Safety - adverse event rate | through study completion, an average of 12 weeks
  Proportion of patient experiencing an adverse event associated with device use

OTHER OUTCOMES:
pain change | 2, 4, 9 and 12 after treatment start
  Pain measured with Visual Analog Scale (VAS) (0-100 mm) at 2, 4, 9 and 12 weeks after treatment start to assess short-term and long-term pain management compared to baseline
Joint stiffness and function | 2, 4, 6 ans 12 weeks after treatment start
  Joint stiffness and function measured with KOOS - Knee Injury and Osteoarthritis Outcome Score [that consists of five sub-scales: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items)]; Quality of Life (four items) for a totoal of 42 items. KOOS max score is 100 and minimum is 0 where zero representing extreme knee problems and 100 representing no knee problem. KOOS will be assessed at 2, 4, 6 and at 12 weeks and compared to baseline.
Patient overall status change | 2, 4, 6 ans 12 weeks after treatment start
  Patient ratings of overall improvement, assessed by QoL (SF-12): The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The SF-12 uses 12 items and scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. SF-12 will be assessed at 2, 4, 6 weeks and at 12 weeks and compared to baseline
Physical function | 2, 4, 6 and 12 weeks after treatment start
  Physical functional test (30 seconds chair-rise test) assessed at 2, 4, 6 and at 12 weeks, compared to baseline.
pain change | 18 weeks after treatment start
  pain measured with Visual Analog Scale (VAS) (0-100 mm) to assess post study pain change (for those patients who did not initiate a new treatment for knee osteoarthritis pain after week 12 and within week 18)
rate of patients needed new treatment | 18 weeks after treatment start
  Patients will be asked through a questionnaire whether any new treatment and in case which one (pharmacological, physiotherapic etc) was needed to manage knee osteoarthritis pain since12 weeks after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Bonthoux, Physiotherap, Principal Investigator — Cabinet d'Ostéopathie
Locations (7):
- France (2):
  - Cabinet d'Ostéopathie, Grésy-sur-Aix
  - Cabinet Allaire, Le Havre
- Italy (4):
  - Casertafisio, Caserta
  - Fisioterapia Carioni, Milan
  - Fisioterapia EUR, Roma
  - Fisioterapia Gardenie, Roma
- Indergaard Physiotherapy, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No